CLINICAL TRIAL: NCT03454438
Title: Strategies to Improve Appropriate Referral to Rheumatologists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: The JOINT referral study
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Rheumatic Disease; Arthralgia
Keywords: Referral; Primary care; Rheumatologist
MeSH Terms: conditions — Rheumatic Diseases; Arthralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Algorithm (Experimental): Use of electronic structured referral sheets using the algorithms for rheumatoid arthritis, axial spondyloarthritis and psoriatic arthritis.
  Interventions: Procedure: Referral strategies
- Triage (Experimental): Triage by rheumatologist in a primary care setting.
  Interventions: Procedure: Referral strategies
- Usual care (No Intervention): Control group consisting of usual care.

INTERVENTIONS:
Procedure: Referral strategies — Two referral strategies will be compared to usual care, i.e. the control group. Patients will be followed for one year.
  Arms: Algorithm; Triage

SUMMARY:
The aim of this cluster randomized controlled trial is to improve the number of effectively referred patients with IRD to the rheumatology outpatient clinic with either use of validated referral pro formas or triage of IRD by specialists in a primary care setting compared to usual care. In addition, the investigators want to provide tools for the general practitioner to recognise IRD and improve early referral of patients with IRD, and a cost-effectiveness analysis will be performed to evaluate the decreasing effect on health-care cost.

DETAILED DESCRIPTION:
Rationale: Currently, only 22% of all patients referred to the rheumatologist by primary care are diagnosed with an inflammatory rheumatic disease (IRD). Previous research has shown that structured referral sheets and community-based specialist service improve appropriateness of referrals.

Objective: The aim of this study is to improve the number of effectively referred patients with IRD to the rheumatology outpatient clinic with either use of validated referral pro formas or triage of IRD by specialists in a primary care setting compared to usual care. In addition, the investigators want to provide tools for the general practitioner to recognise IRD and improve early referral of patients with IRD, and a cost-effectiveness analysis will be performed to evaluate the decreasing effect on health-care cost.

Study design: Cluster randomized trial with randomization of general practitioner clinics.

Study population: Primary care patients of 18 years or older who are suspected of an IRD and considered by a GP for referral to a rheumatologist.

Intervention: One group of GPs will use a standardized referral strategy for IRD, another group will consist of triage by a rheumatologist in the local primary care clinic, the third group is usual care.

Main study parameters/endpoints: Percentage of patients diagnosed with an IRD by a rheumatologists after 12 months. In addition, cost effectiveness, quality of life, work participation and health care costs at baseline and after 12 months.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no additional risk to participating patients. Patients might benefit from early referral since the referral pro formas point out important aspects of IRD that are frequently overlooked. Patients will be requested to fill in three online questionnaires related to quality of life, work participation and socio-economic costs. There are no additional visits, physical examinations or other tests.

ELIGIBILITY:
Inclusion Criteria:

* A primary care patient who is referred by the GP to the rheumatology outpatient clinic
* Subject must be able to understand and communicate with the rheumatologist
* Participant must give a written signed and dated informed consent before enrolment.

Exclusion Criteria:

* Limited understanding of the Dutch language.
* Legally incapable or vulnerable subject as described in the Medical Research with Human Subjects Act (WMO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of appropriate referred patients | 12 months
  Percentage of appropriate referred patients as proportion of all patients referred to the rheumatologist by the general practitioner (GP). Appropriate referred defined as patient diagnosed with an inflammatory rheumatic disease (IRD) as assessed by a rheumatologist, with an IRD as final diagnosis.

SECONDARY OUTCOMES:
EuroQoL Health questionnaire | 12 months
  The standard analysis for health-related quality of life in cost-effectiveness research, tool in determining Quality adjusted life years (QALYs).
iMTA Medical Consumption Questionnaire | 12 months
  Collects information on non-disease specific health-care consumption.
iMTA Productivity Cost Questionnaire | 12 months
  Measurement of productivity loss and work participation.
Health-care costs | 12 months
  Amount of outpatient clinic visits (visits to medical specialist, supporting staff, other staff), diagnostics (laboratory analyses, imaging), therapy (medication, medical procedures, over the counter medication), general practitioner consultation, medication use prescribed by general practitioner.

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Weel-Koenders, Principal Investigator — Maasstad Hospital
Locations (1):
- Maasstad Hospital, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] van Delft ETAM, Barreto DL, van der Helm-van Mil AHM, Alves C, Hazes JMW, Kuijper TM, Weel-Koenders AEAM. Diagnostic Performance and Clinical Utility of Referral Rules to Identify Primary Care Patients at Risk of an Inflammatory Rheumatic Disease. Arthritis Care Res (Hoboken). 2022 Dec;74(12):2100-2107. doi: 10.1002/acr.24789. Epub 2022 Jul 31. PMID 34553506